CLINICAL TRIAL: NCT07284563
Title: Evaluation of Ultralow Dose PET Imaging for Detecting 18F-NaF Uptake
Brief Title: Ultralow Dose PET Imaging for 18F-NaF Uptake
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akiva Mintz (Other)
Responsible Party: Sponsor-Investigator, Akiva Mintz, Executive Director, Nuclear Imaging Institute
Organization: Nuclear Imaging Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NII-0003-NaF
Record Dates: First submitted 2025-12-08; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer; Bone Alteration; Bone and Joint Cancer; Bone and Joint Infection; Arthritis
Keywords: PET; PET/CT; low dose; nuclear imaging; sodium fluoride; bone
MeSH Terms: conditions — Arthritis | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, single-center imaging study designed to evaluate the optimal timing and reconstruction parameters for ultralow dose 18F-NaF imaging using a long axial field-of-view (LAFOV) PET scanner.
  The study aims to determine whether normal and diseased tissue can be accurately visualized at significantly lower radiotracer doses, while optimizing scan duration and reconstruction methods to maintain diagnostic performance.
  A total of 200 participants will be enrolled in a single cohort, including healthy volunteers and individuals with suspected or confirmed increased bone turnover that is found in diseases such as cancer, trauma, infection, arthritis, and other benign diseases of bone. The inclusion of both healthy and diseased subjects allows for a comprehensive evaluation of normal organ uptake patterns, which is the primary objective of the study. Participants will undergo a single PET scan session per an enrollment, and be eligible for re-enrollment after 6 m
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ultralow dose 18F-NaF imaging group (Other): Participants will be enrolled for an ultralow dose PET scan to evaluate image quality and optimize timing and reconstruction after reducing radiation doses 10-100 fold. Participants will be injected with a very small amount of radiotracer and imaged on a PET scanner for up to 3 hours
  Interventions: Drug: 18F-NaF

INTERVENTIONS:
Drug: 18F-NaF — Participants will be injected with 18F-NaF and imaged for up to 3 hours on a PET scanner
  Other Names: CT scan; PET scan; blood collection

SUMMARY:
The goal of this clinical trial is to evaluate an investigational ultralow dose positron emission tomography (PET imaging) technique for increased bone turnover that is found in diseases such as cancer, trauma, infection, arthritis, and other benign diseases of bone detection and monitoring. The main question it aims to answer is:

Can the investigators optimize the timing, scan duration, and image reconstruction to reduce the radiation dose 10-100 fold of the current clinical standard? Participants will be injected with a radioactive tracer called Fluorine-18 (18F)-sodium fluoride (NaF) and be imaged on a new type of high sensitivity PET scanner for up to 3 hours.

DETAILED DESCRIPTION:
This research study aims to evaluate an investigational ultralow dose PET imaging technique for increased bone turnover that is found in diseases such as cancer, trauma, infection, arthritis, and other benign diseases of bone detection and monitoring. "Investigational" means that the procedure or drug being studied is not yet approved by the FDA for the specific use being tested in this research. The PET imaging technique used in this study is considered investigational because it is being tested at an ultralow radiation dose that has not yet been approved for clinical use. The radiotracer, 18F-NaF, is FDA-approved for detecting prostate cancer at standard doses.

18F-NaF is often found to be taken up at higher levels in increased bone turnover that is found in diseases such as cancer, trauma, infection, arthritis, and other benign diseases of bone. In this study, investigators will use a very small amount of this tracer (less than 1/20th of the standard dose) along with advanced PET imaging technology to see if it is possible to create clear images while using much less radiation. This study aims to develop a safer imaging technique that could potentially be used more frequently for screening and monitoring increased bone turnover that is found in diseases such as cancer, trauma, infection, arthritis, and other benign diseases of bone.

Investigators will enroll individuals with and without increased bone turnover that is found in diseases such as cancer, trauma, infection, arthritis, and other benign diseases of bone to evaluate how ultralow dose PET imaging detects 18F-NaF uptake in different type of tissue.

Approximately 200 people will be enrolled in this study at the Nuclear Imaging Institute.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Ability to provide informed consent and comply with study procedures.
* For female participants: Must not be pregnant or breastfeeding; Negative pregnancy test required for women of childbearing potential.

Exclusion Criteria:

* Participants who have exceeded NRC regulation for annual radiation exposure from prior research-related scans, including this study (50 millisievert [mSv] total).
* More than four prior enrollments in this study.
* Participants with severe claustrophobia, chronic pain, or musculoskeletal conditions that prevent completion of the PET scan
* Medication & Prior Treatment Exclusions
* Concurrent treatments that may interfere with radiotracer uptake as determined by the Principle Investigator.
* Pregnant or breastfeeding individuals (negative pregnancy test required)
* Inability to provide informed consent
* Any condition that, in the investigator's judgment, may compromise participant safety or study integrity.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Signal-to-Noise Ratio (SNR) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Measurement of signal-to-noise ratio for image quality assessment across different scan durations, reconstruction techniques, and AI-enhanced image reconstructions. Unit of Measure: SNR (unitless, numeric ratio)
Contrast-to-Noise Ratio (CNR) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Measurement of contrast-to-noise ratio for image quality assessment across different scan durations, reconstruction techniques, and AI-enhanced image reconstructions. Unit of Measure: CNR (unitless, numeric ratio)
Coefficient of Variation (COV) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Measurement of the coefficient of variation in selected regions for evaluating image consistency across different scan durations, reconstruction techniques, and AI-enhanced image reconstructions. Unit of Measure: Percentage (%)
Spatial Resolution (Full Width at Half Maximum - FWHM) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Assessment of spatial resolution using full width at half maximum (FWHM) across different scan durations, reconstruction techniques, and AI-enhanced image reconstructions. Unit of Measure: Millimeters (mm)
Target-to-Background Ratio (TBR) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Assessment of target-to-background ratio for evaluating PSMA-expressing tissue contrast across different scan durations, reconstruction techniques, and AI-enhanced image reconstructions. Unit of Measure: Ratio (unitless numeric ratio)
Qualitative Image Quality Score (Likert Scale) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Independent qualitative evaluation of overall image quality, lesion detectability, image noise, and artifacts by nuclear medicine physicians, assessed using a 5-point Likert scale. Unit of Measure: Score on Likert Scale (1-5; 1 = worst, 5 = best)
Inter-reader Agreement (Weighted Kappa Statistics) | Evaluated annually (once per year), based on pooled images acquired during the preceding 12-month period.
  Measurement of agreement among readers evaluating qualitative image quality scores, analyzed using weighted kappa statistics. Unit of Measure: Weighted kappa statistic (numeric value ranging from 0 to 1, 0 = no agreement, 1 = perfect agreement)

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear Imaging Institute, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided